CLINICAL TRIAL: NCT03585556
Title: A Phase 1 Proof of Concept Study Evaluating Intravitreal AAVCAGsCD59 for the Treatment of Wet Age-Related Macular Degeneration (AMD)
Brief Title: AAVCAGsCD59 for the Treatment of Wet AMD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 81201887MDG1002; HMR-1002 (Other: Janssen Research & Development, LLC); 81201887MDG1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-07-01; First posted 2018-07-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Wet Age-related Macular Degeneration
Keywords: Wet Age-related Macular Degeneration; Gene therapy; Wet AMD
MeSH Terms: interventions — Bevacizumab; Ranibizumab; aflibercept; Prednisolone; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: All patients with treatment naive, new onset wet AMD will be treated with an intravitreal anti-VEGF at Day 0 followed by intravitreal AAVCAGsCD59 at Day 7. Patients will be followed for 12 months and treated with additional anti-VEGF monthly as needed if recurrent disease is identified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AAVCAGsCD59 Treated Arm (Experimental): An anti-VEGF injection will be given at Day 0 followed by an intravitreal injection of AAVCAGsCD59 at Day 7. All eyes will then be treated with intravitreal anti-VEGF monthly as needed based on disease activity.
  Interventions: Drug: Intravitreal anti-VEGF; Biological: Intravitreal AAVCAGsCD59; Drug: Oral prednisolone

INTERVENTIONS:
Drug: Intravitreal anti-VEGF — Intravitreal injection of anti-VEGF at Day 0 then monthly as needed
  Other Names: Bevacizumab (Avastin); Ranibizumab (Lucentis); Aflibercept (Eylea)
Biological: Intravitreal AAVCAGsCD59 — An intravitreal injection of AAVCAGsCD59 will occur at Day 7 once
  Other Names: HMR59
Drug: Oral prednisolone — A 7 day tapering dose of oral prednisone will be taken at Day 30 by all patients
  Other Names: oral corticosteroid

SUMMARY:
Patients with treatment naive wet AMD will receive an intravitreal anti-VEGF injection at Day 0 followed by an intravitreal injection of AAVCAGsCD59 at Day 7. Patients will be followed monthly through Month 12 and receive an intravitreal anti-VEGF injection as needed based on an increase in central subfoveal thickness (CST) of >50 micrometers on OCT from Day 0, new subretinal hemorrhage on clinical exam, and/or loss of 10 or more ETDRS letters from the previous month exam.

DETAILED DESCRIPTION:
This is a Phase 1, multi-center, open label study to assess the efficacy and safety of two doses of the adeno-associated viral vector serotype 2 (AAVCAGsCD59) expressing sCD59 administered via intravitreal injection seven days after a single intravitreal injection of anti-VEGF. All patients considered for enrollment in this study must have treatment naive wet AMD, adequate pupillary dilation to permit a thorough ocular exam, and best corrected distance visual acuity in the study eye of 20/25 to 20/400 using the Snellen eye chart.

Written informed consent will be obtained from each study patient prior to his/her participation in any study related procedures. Screening will determine patient eligibility for the study according to written inclusion and exclusion criteria, which include both general medical and AMD-specific criteria. Patients will be enrolled into the study upon verification that they fulfill all eligibility criteria and after completion of all screening assessments.

This study consists of a screening and injection of anti-VEGF (Day 0), injection of AAVCAGsCD59 (Day 7), and a monthly follow-up period (Month 1 through Month 12) where enrolled patients are treated as needed with intravitreal anti-VEGF based on an increase in central subfoveal thickness of >50 micrometers on OCT from Day 0, new subretinal hemorrhage, a decrease in > or equal to 10 ETDRS letters from the previous exam, or as needed based on the treating clinician. The purpose of the study is to evaluate the number of anti-VEGF injections that are required after a single intravitreal injection of AAVCAGsCD59 at a dose of 3.56x10e11vg for subjects 1-22 and 1.071x10e12vg for subjects 23-25 is administered on Day 7. Anti-VEGF will be injected at Day 0 to treat the CNV per standard of care and enable the AAVCAGsCD59 adequate time (up to two weeks) to enter the ganglion cells in the retina and start producing the transgene product, sCD59. Up to twenty-five (25) patients will be enrolled at to 2 clinical sites in this study. A long-term follow-up safety exam will occur at Month 24.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women 50 years of age or older.
2. Treatment naive Wet AMD with no evidence of subretinal fibrosis under the fovea.
3. Presence of intraretinal and/or subretinal fluid on OCT.
4. Best corrected visual acuity (BCVA) Snellen equivalent 20/25 to 20/400 in the study eye using ETDRS charts at a starting distance of 4m.
5. Adequate pupillary dilation to permit ocular examination and testing.
6. Ability and willingness to return for all scheduled visits and assessments.
7. Understand and comply with the clinical protocol and provide written informed consent prior to any study-related procedure.
8. All fertile men must be willing to use barrier contraception during the study.
9. Women of childbearing potential must have a negative pregnancy test and agree to use effective contraception for the duration of the trial. A woman of childbearing potential is defined as any female who has had menses within the last two years or has not undergone a hysterectomy or surgical sterilization.

Exclusion Criteria:

1. Wet AMD secondary to non-AMD etiologies.
2. Subretinal hemorrhage that interferes with the ability to adequately measure visual acuity or follow retinal or subretinal fluid collection on OCT.
3. Serous pigment epithelial detachment (PED) that is >50% of the CNV lesion, >400µm in any diameter, or presence of a RPE tear.
4. Presence of polypoidal choroidal vasculopathy (PCV), retinal angiomatous proliferation (RAP), central serous retinopathy, or symptomatic vitreomacular adhesion.
5. Previous macular laser photocoagulation for CNV, photodynamic therapy (PDT), ocular radiation, or subretinal surgery for CNV in the study eye.
6. History of conditions in the study eye which might alter visual acuity or interfere with study testing including clinically significant macular edema, central retinal vein occlusion, macular branch retinal vein occlusion, and optic neuropathy.
7. Active uncontrolled glaucoma with IOP>30 mmHg despite treatment with glaucoma medications, cup-to-disc ratio of >0.9, visual field defects secondary to glaucoma that involve the macula, and optic atrophy from glaucoma.
8. Likely candidate for intraocular surgery (including cataract surgery) in the study eye during the clinical trial.
9. Acute or chronic infection in the study eye.
10. History of uveitis unrelated to eye surgery in the study eye or opposite eye requiring treatment with topical corticosteroids or systemic immunosuppression within 24 months of enrollment.
11. Any contraindication to intravitreal injection.
12. Use intravitreal (study eye) corticosteroids within 3 months prior to screening.
13. Any of the following underlying systemic diseases:

    * Unstable or severe cardiovascular disease, e.g., congestive heart failure (New York Heart Association Functional class III or IV), myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina, or critical limb ischemia;
    * Cerebrovascular disease within 12 months prior to Screening that impairs the patient's ability to participate in the clinical trial;
    * Dementia or neurodegenerative disease (e.g., Alzheimer's disease, Parkinson's disease) of a level that prevents adequate evaluation of the subject during the study;
    * Has an active malignancy or is currently undergoing treatment for an active malignancy at Screening, or has a history of malignancy that precludes completion of this 12-month study;
    * Immunocompromised conditions and/or need for immunosuppressive therapy
14. Any significant poorly controlled illness that would preclude study compliance and follow-up
15. Current or prior use of any medication known to be toxic to the retina or optic nerve including, but not limited, to chloroquine/hydrochloroquine, deferoxamine, phenothiazines and ethambutol
16. Previous treatment with any ocular or systemic gene transfer product
17. Received any investigational product within 120 days prior to screening
18. Any psychological, familial, sociological, geographical, or other condition that would preclude study compliance and follow-up

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Number of intravitreal anti-VEGF injections | 12 months
  Measure the number of intravitreal anti VEGF injections from Month 1 through Month 12 following an intravitreal injection of AAVCAGsCD59 at Day 7

SECONDARY OUTCOMES:
Number of patients with change in vision of ≥ 15 letters | 12 months
  Evaluate the change in vision in eyes receiving intravitreal AAVCAGsCD59 in conjunction with anti VEGF for new onset wet AMD
Number of patients with inflammation, endophthalmitis, IOP>30, retinal detachment, cataract, and systemic adverse events | 24 months
  Evaluate SAEs associated with the use of intravitreal AAVCAGsCD59

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Vitreo-Retina Associates, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No